CLINICAL TRIAL: NCT04546230
Title: Low-Thoracic Epidural Anesthesia For Laparoscopic Nephrectomy In Adult Patients.
Brief Title: Low-Thoracic Epidural Anesthesia For Laparoscopic Nephrectomy.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nazmy Edward Seif (Other)
Responsible Party: Sponsor-Investigator, Nazmy Edward Seif, Clinical Professor, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: LTEALN
Record Dates: First submitted 2020-09-06; First posted 2020-09-11 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Laparoscopic; Nephrectomy; Anesthesia; Epidural
Keywords: Epidural Anesthesia; Low-thoracic; Laparoscopic nephrectomy
MeSH Terms: interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E group (Experimental): Low-Thoracic Epidural Anesthesia
  Interventions: Procedure: Low-Thoracic Epidural Anesthesia
- G group (Active Comparator): General Anesthesia
  Interventions: Procedure: General Anesthesia

INTERVENTIONS:
Procedure: Low-Thoracic Epidural Anesthesia — Under aseptic conditions and local anesthesia, an epidural catheter will be inserted using the "Prefix Epidural Anesthesia Tray" with an 18 G Tuohy needle & a 20 G catheter at the T7-8 or T8-9 intervertebral space. The epidural catheter will be threaded leaving 3 cm within the epidural space and tapped in place.
  Using a mixed preparation of isobaric Bupivacaine 0.5% with Fentanyl 2 μg per ml volume, a bolus dose of 5-10 ml will then be given via the epidural catheter, followed by 5-10 ml/hr as a continuous infusion to be started 1 hour later & continued throughout the procedure.
  Arms: E group
Procedure: General Anesthesia — General anaesthesia will be induced with intra-venous administration of Fentanyl (2 μg/kg), Propofol (2 mg/kg), Atracurium (0.5 mg/kg) and Lidocaine (1 mg/kg). After tracheal intubation, balanced anaesthesia will be maintained with isoflurane in oxygen & infusion of atracurium at a rate of 0.5 mg/kg/hr; and mechanical ventilation will be provided.
  Arms: G group

SUMMARY:
Laparoscopic nephrectomy is a surgical technique to excise a diseased kidney. It's a minimally invasive technique, so when compared to open surgery, it can mean significantly less post-operative pain, shorter hospital stay, earlier return to work and daily life activities, a more favourable cosmetic result and outcomes similar to that of open surgery.

Recently, advanced laparoscopic surgery has targeted older and high risk patients for general anesthesia; in these patients, regional anesthesia offers several advantages with improved patient satisfaction. Compared with alternative anesthetic techniques, epidural anesthesia may reduce the risks of venous thromboembolism, myocardial infarction, bleeding complications, pneumonia, respiratory depression and renal failure.

The aim of this study is to compare the conventional general anesthetic technique to the regional anesthesia for laparoscopic nephrectomy, in modified lateral decubitus position using low-pressure pneumoperitoneum.

ELIGIBILITY:
Inclusion Criteria:

* ASA I - II.
* Adult patients scheduled for laparoscopic nephrectomy.

Exclusion Criteria:

* Patient refusal.
* Contraindication to regional anesthesia (e.g., coagulopathy, site infection).
* Allergy to local anesthetics.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-09-19 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overall patient satisfaction. | 24 hours
  The overall degree of patients' satisfaction will be assessed using a "5-point patient satisfaction rating scale" according to Likert scale [where: very unsatisfied=1/5, unsatisfied=2/5, neutral=3/5, satisfied=4/5, and very satisfied=5/5].

CONTACTS AND LOCATIONS:
Overall Officials: Nazmy S Michael, MD, Principal Investigator — Kasr Al-Ainy Hospital, Faculty of Medicine, Cairo University; Atef K Salama, MD, Study Director — Kasr Al-Ainy Hospital, Faculty of Medicine, Cairo University
Locations (1):
- Cairo University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided